CLINICAL TRIAL: NCT00712894
Title: Reversal of No-reflow/Slow-flow During Percutaneous Coronary Intervention in Patients With Acute Myocardial Infarction--a Prospective Randomized Study Comparing Intracoronary Infusion of Diltiazem, Verapamil and Nitroglycerin
Brief Title: Effects of Different Vasodilators on Coronary No-reflow During primAry percuTaneous Coronary intErvention in Patients With Acute Myocardial Infarction
Acronym: EDUCATE-AMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ge Junbo, Director of Cardiology Department, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zhongshan 2006-70
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Acute Myocardial Infarction; Percutaneous Coronary Intervention
Keywords: Acute myocardial infarction; Percutaneous coronary intervention; No-reflow phenomenon; Vasodilator agents
MeSH Terms: conditions — No-Reflow Phenomenon | interventions — Diltiazem; Verapamil; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- D (Experimental): If no-reflow/slow-flow phenomenon was observed post-PCI, intracoronary infusion of diltiazem via an infusion microcatheter distal to the angioplasty site was performed.
  Interventions: Drug: Diltiazem
- V (Active Comparator): If no-reflow/slow-flow phenomenon was observed post-PCI, intracoronary infusion of verapamil via an infusion microcatheter distal to the angioplasty site was performed.
  Interventions: Drug: Verapamil
- N (Active Comparator): If no-reflow/slow-flow phenomenon was observed post-PCI, intracoronary infusion of nitroglycerin via an infusion microcatheter distal to the angioplasty site was performed.
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Diltiazem — Intracoronary Infusion 400-2000ug
  Arms: D
Drug: Verapamil — Intracoronary Infusion 200-1000ug
  Arms: V
Drug: Nitroglycerin — Intracoronary Infusion 200-1000ug
  Arms: N

SUMMARY:
The purpose of this study is to evaluate the efficacy of three different vasodilators including diltiazem, verapamil and nitroglycerin for reversal of no-reflow/slow-flow during direct percutaneous coronary intervention for acute myocardial infarction.

DETAILED DESCRIPTION:
No-reflow/slow-flow is a frequent observation during direct PCI for AMI and associated with a poor clinical outcome. The present pharmacological management involves the use of different vasodilators including nitrates, verapamil, adenosine and nicorandil. But no randomized trial has been conducted to assess any of these agents, or to determine the appropriate dosage. This prospective randomized study aimed to confirm favorable effects of diltiazem on no-reflow/slow-flow during direct PCI for AMI compared with verapamil and nitroglycerin.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myocardial infarction
* Vessel TIMI flow < grade Ⅲ post-PCI

Exclusion Criteria:

* Heart failure of New York Heart Association (NYHA) class Ⅲ to class Ⅳ
* Sick sinus syndrome
* Atrioventricular block (grade Ⅱ and above)
* SBP ≤ 90mmHg or cardiogenic shock
* Heart Rate ≤60 bpm
* Pregnancy
* Renal or hepatic failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Vessel flow using TIMI flow grade and TIMI frame count | post-PCI

SECONDARY OUTCOMES:
major adverse cardiovascular events (MACE) | within the first 30 days after PCI
Left ventricular ejection fraction (LVEF) through echocardiography | at 1 and 30 days post-PCI
NT-proBNP levels | at 1 and 30 days post-PCI
incidence of complete ST-segment resolution | 3 hours after PCI
peak troponin T level | 24 hours after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Huang D, Qian J, Ge L, Jin X, Jin H, Ma J, Liu Z, Zhang F, Dong L, Wang X, Yao K, Ge J. REstoration of COronary flow in patients with no-reflow after primary coronary interVEntion of acute myocaRdial infarction (RECOVER). Am Heart J. 2012 Sep;164(3):394-401. doi: 10.1016/j.ahj.2012.06.015. PMID 22980307